CLINICAL TRIAL: NCT01348022
Title: Prospective Evaluation of Outcomes of Everolimus-Eluting Stent (XIENCE V) Implantation for Unprotected Left Main Coronary Artery Stenosis: Multicenter Trial
Brief Title: Evaluation of Outcomes of EES Implantation for Unprotected Left Main Coronary Artery Stenosis (PRE-COMBAT 2)
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D., Ph.D.,Professor of Medicine Asan Medical Center, University of Ulsan, College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: 2009-0361
Record Dates: First submitted 2011-04-22; First posted 2011-05-05 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Xience V stent: unprotected Left Main Coronary Artery stenting treated with Xience V stent

SUMMARY:
This study is a multicenter, open label, prospective, single arm trial

Single arm group; following angiography, eligible patients with unprotected LMCA stenosis >50% by visual estimation, which is equally treatable by the both treatment strategy (EES stenting or CABG), will be treated with EES

DETAILED DESCRIPTION:
The primary objective of the PRECOMBAT-2 trial is to establish the safety and effectiveness of coronary stenting with the everolimus-eluting Xience V stent (EES) compared with the historical control (PRE-COMBAT-1) of bypass surgery and sirolimus-eluting stent (SES) for the treatment of an unprotected LMCA stenosis. The primary alternative hypothesis is that the experimental starategy (coronary stenting with the everolimus-eluting stents) is not inferior to the standard strategy (CABG) or SES.

All consecutive patients with unprotected LMCA diseases at participating centers, who are treated with Xience V stent, will be evaluated for the entry into the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years of age.
2. Significant de novo left main stenosis (>50% by visual estimation) with or without any additional target lesions (>70% by visual estimation)
3. Left main lesion and lesions outside LMCA (if present) potentially equally treatable with coronary stenting and CABG
4. Patients with stable (CCS class 1 to 4) or acute coronary syndromes (unstable angina pectoris Braunwald class IB, IC, IIB, IIC, IIIB, IIIC or NSTEMI) or patients with atypical chest pain or without symptoms but having documented myocardial ischemia
5. The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications:

   * Heparin
   * Aspirin
   * Both Clopidogrel and TIclopidine
   * Everolimus, paclitaxel, ABT 578
   * Stainless steel and/or
   * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
2. Systemic (intravenous) Everolimus, paclitaxel or ABT-578 use within 12 months.
3. Any previous PCI within 1 year
4. Previous bypass surgery
5. Any previous PCI of a LMCA or ostial left circumflex artery or ostial left anterior descending artery lesion within 1 year
6. Intention to treat more than one totally occluded major epicardial vessel
7. Acute MI patients within 1 week
8. Patients with EF<30%.
9. Patients with cardiogenic shock
10. Any disabled stroke with neurological deficit or any cerebrovascular accident within 6 months
11. Creatinine level 2.0mg/dL or dependence on dialysis.
12. Severe hepatic dysfunction (AST and ALT 3 times upper normal reference values).
13. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
14. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
15. Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
16. An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 1 year post enrollment.
17. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
18. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
19. Subject unable or unwilling to follow-up with visits required by protocol
20. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery disease requiring drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
MACCE free survival | at 2 year
  Death (all-cause mortality) Cerebrovascular accident Non-fatal myocardial infarction (Q wave and non-Q wave) Ischemia-driven target vessel revascularization either percutaneous or surgical treatment

SECONDARY OUTCOMES:
Death(all cause and cardiac) | 5 years
Myocardial Infarction | 5 years
Cerebrovascular accident | 5 years
Target vessel revascularization | 5 years
Target lesion revascularization | 5 years
Stent thrombosis | 5 years
Binary restenosis in both in-stent and in-segment | 9 months
  angiographic follow-up
Late luminal loss in both in-stent and in-segment | 9 months
  angiographic follow-up
pattern of restenosis | 9 months
  angiographic follow-up
Angina status | 5 years
Re-hospitalization with a cardiac cause | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (21):
- South Korea (21):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Kwangju Christian Hospital, Kwangju
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Veterans Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Derived] Kim YH, Park DW, Ahn JM, Yun SC, Song HG, Lee JY, Kim WJ, Kang SJ, Lee SW, Lee CW, Park SW, Jang Y, Jeong MH, Kim HS, Hur SH, Rha SW, Lim DS, Her SH, Seung KB, Seong IW, Park SJ; PRECOMBAT-2 Investigators. Everolimus-eluting stent implantation for unprotected left main coronary artery stenosis. The PRECOMBAT-2 (Premier of Randomized Comparison of Bypass Surgery versus Angioplasty Using Sirolimus-Eluting Stent in Patients with Left Main Coronary Artery Disease) study. JACC Cardiovasc Interv. 2012 Jul;5(7):708-17. doi: 10.1016/j.jcin.2012.05.002. PMID 22814775